CLINICAL TRIAL: NCT00909844
Title: Follow-up of the Phase III, Multicentre, Non Comparative, One Single Group, Open Study to Assess the Long-term Efficacy and Tolerability of Pamoate of Triptorelin 11.25 mg in Children With Precocious Puberty
Brief Title: Effects of Triptorelin Pamoate in Children With Precocious Puberty - Follow up Study
Acronym: DECAPUB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-54-52014-159; 2008-000565-39 (EudraCT Number)
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Precocious Puberty
MeSH Terms: conditions — Puberty, Precocious | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triptorelin (Experimental)
  Interventions: Drug: Triptorelin (I.N.N.)

INTERVENTIONS:
Drug: Triptorelin (I.N.N.) — Decapeptyl® SR 11.25mg

SUMMARY:
The purpose of the protocol is to assess the efficacy of triptorelin 11.25 mg with respect to the proportion of children who maintain a regression or stabilisation of sexual maturity until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* The child must have completed study 2-54-52014-143
* The child must have an effective response to 2 injections of triptorelin 11.25 mg according to investigator's evaluation with no significant treatment side effects

Exclusion Criteria:

* The patient has a known hypersensitivity to any of the test materials or related compounds
* The patient is unable or unwilling to comply fully with the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-04; Primary Completion 2015-04 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- France (10):
  - Hôpital Hôtel Dieu (CHU), Angers
  - Medical Centre, Bordeaux
  - Hôpital Flaubert, Le Havre
  - Hôpital Archet II, Nice
  - Hôpital Robert Debré, Paris
  - American Memorial Hospital, Reims
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Hautepierre, Strasbourg
  - Hôpital de la Gespe, Tarbes
  - Hôpital des Enfants, Toulouse

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed as a multicentre study and included 10 investigational sites in France. This follow up study was to start on the day of the last visit (Month 6) of the phase III 2-54-52014-143 study and was to end when the Investigator judged that the patient had completed his/her treatment, i.e. at around 11 years in girls and 13 in boys.
Pre-assignment Details: A maximum of 35 patients could be included in this study (i.e. the number of patients who had completed the phase III 2-54-52014-143 study). A total of 35 patients were screened and enrolled in this current study (2-54-52014-159).
Groups:
- Triptorelin Pamoate 11.25 mg: 11.25 mg triptorelin pamoate (prolonged release formulation) was administered via intramuscular (i.m.) injection once every 3 months from Baseline until end of the study treatment.
Period: Overall Study
Arm/Group | Triptorelin Pamoate 11.25 mg
Started | 35
Completed | 31
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for Intention-To-Treat Population (ITT) population, consisting of all enrolled patients who received at least one injection of study treatment in this follow up study. These data were not re-collected at the start of the current study and are derived from data collected at Baseline of study 2-54-52014-143.
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.73 (1.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 1
Weight at Pretreatment [Mean (Standard Deviation); unit: kilogram (kg)] | 32.4 (6.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Children With a Stabilisation or Regression of Tanner Pubertal Stage at the End of the Study (Final Visit), Compared to Pretreatment (Month -6) and Baseline (Month 0)
Description: The primary objective was to assess efficacy of triptorelin pamoate 11.25 mg with respect to percentage of children maintaining a regression or stabilisation of sexual maturity (based on Tanner breast [girls] or genital [boys] pubertal stage) until end of study. Study treatment lasted until end of the therapeutic period; visits for Months 36 and 48 were optional since a child may have already finished the study at a prior visit. The Final Visit only occurred if the child did not end the study by a complete visit such as at Months 24, 36 or 48. Results are presented only for percentage of girls with regression or stabilisation of Tanner breast pubertal stage (n=34). Since only one boy was included in the study, results for this outcome measure were listed only and no statistical analysis was performed. Please also note additional post-hoc analysis for regression or stabilisation of Tanner breast pubertal stage which applied the variable Last Visit on Treatment instead of Final Visit.
Time Frame: Months 12, 24, 36, 48 and Final Visit (if applicable; up to 63 months)
Population: Analysis performed on female patients in the ITT population, consisting of all enrolled female patients who received at least one injection of study treatment in this follow up study.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 34
percentage of patients
  Compared to Pretreatment (Month -6) | 61.8 [43.56 to 77.83]
  Compared to Baseline (Month 0) | 52.9 [35.13 to 70.22]

2. Secondary Outcome: Percentage of Patients With a Suppressed Luteinizing Hormone (LH) Response to Gonadotropin-Releasing Hormone (GnRH) Test
Description: A suppressed LH response to the GnRH test was defined as a stimulated peak of LH ≤3 international units per litre (IU/L). Percentage of patients who had a suppressed LH response to the GnRH test is reported. It should be noted that almost no hormonal data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0 and 36
Population: Analysis performed on the ITT population, consisting of all enrolled patients who received at least one injection of study treatment in this follow up study. Only patients with data available at the timepoint of testing are reported.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Triptorelin Pamoate 11.25 mg: 11.25 mg triptorelin pamoate (prolonged release formulation) was administered via i.m. injection once every 3 months from Baseline until end of the study treatment.
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
percentage of patients
  Pretreatment (Month -6) | 0 [NA to NA] — At Pretreatment, 0 patients had suppressed LH response to the GnRH test so 95% confidence interval is not applicable.
  Baseline (Month 0) | 91.4 [76.94 to 98.20]
  Month 36: number analyzed (Participants) | 1
  Month 36 | 100 [2.50 to 100.00]

3. Secondary Outcome: Levels of Oestradiol in Girls or Testosterone in Boys Both Measured by Radioimmunoassay (RIA)
Description: Mean levels of oestradiol in girls or testosterone in boys are reported. It should be noted that almost no hormonal data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0, 12, 36 and Final Visit (up to 63 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picograms per millilitre (pg/mL)
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
picograms per millilitre (pg/mL)
  Oestradiol at Pretreatment (Girls): number analyzed (Participants) | 34
  Oestradiol at Pretreatment (Girls) | 18.59 (9.79)
  Oestradiol at Baseline (Girls): number analyzed (Participants) | 34
  Oestradiol at Baseline (Girls) | 8.71 (4.51)
  Oestradiol at Month 12 (Girls): number analyzed (Participants) | 1
  Oestradiol at Month 12 (Girls) | 2.50 (NA) — No SD is presented since mean value is derived from a single patient
  Oestradiol at Month 36 (Girls): number analyzed (Participants) | 1
  Oestradiol at Month 36 (Girls) | 12.20 (NA) — No SD is presented since mean value is derived from a single patient
  Oestradiol at Final Visit (Girls): number analyzed (Participants) | 1
  Oestradiol at Final Visit (Girls) | 10.00 (NA) — No SD is presented since mean value is derived from a single patient
  Testosterone at Pretreatment (Boy): number analyzed (Participants) | 1
  Testosterone at Pretreatment (Boy) | 6.80 (NA) — No SD is presented since mean value is derived from a single patient
  Testosterone at Baseline (Boy): number analyzed (Participants) | 1
  Testosterone at Baseline (Boy) | 0.56 (NA) — No SD is presented since mean value is derived from a single patient

4. Secondary Outcome: Percentage of Patients With a Suppressed Follicle Stimulating Hormone (FSH) Response to GnRH Test
Description: A suppressed FSH response to the GnRH test was defined as a stimulated peak of FSH ≤3 IU/L. Percentage of patients who had a suppressed FSH response to the GnRH test is reported. It should be noted that almost no hormonal data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0 and 36
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
percentage of patients
  Pretreatment (Month -6) | 0 [NA to NA] — At Pretreatment, 0 patients had suppressed LH response to the GnRH test so 95% confidence interval is not applicable.
  Baseline (Month 0) | 82.9 [66.35 to 93.44]
  Month 36: number analyzed (Participants) | 1
  Month 36 | 0 [NA to NA] — No CIs are presented since percentage value is derived from a single patient

5. Secondary Outcome: Body Mass Index (BMI) for Chronological Age Variation
Description: Mean changes of BMI from Pretreatment and from Baseline are reported. It should be noted that only limited patient data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0, 12, 24, 36, 48 and Final Visit (up to 63 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms per metre squared (kg/m^2)
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
kilograms per metre squared (kg/m^2)
  Change from Pretreatment at Baseline: number analyzed (Participants) | 34
  Change from Pretreatment at Baseline | 0.43 (0.74)
  Change from Pretreatment at Month 12: number analyzed (Participants) | 30
  Change from Pretreatment at Month 12 | 1.60 (1.29)
  Change from Pretreatment at Month 24: number analyzed (Participants) | 16
  Change from Pretreatment at Month 24 | 1.69 (1.60)
  Change from Pretreatment at Month 36: number analyzed (Participants) | 3
  Change from Pretreatment at Month 36 | 1.69 (2.48)
  Change from Pretreatment at Month 48: number analyzed (Participants) | 2
  Change from Pretreatment at Month 48 | 1.06 (1.29)
  Change from Pretreatment at Final Visit: number analyzed (Participants) | 31
  Change from Pretreatment at Final Visit | 2.39 (1.62)
  Change from Baseline at Month 12: number analyzed (Participants) | 29
  Change from Baseline at Month 12 | 1.14 (1.00)
  Change from Baseline at Month 24: number analyzed (Participants) | 14
  Change from Baseline at Month 24 | 1.43 (1.45)
  Change from Baseline at Month 36: number analyzed (Participants) | 3
  Change from Baseline at Month 36 | 1.53 (1.62)
  Change from Baseline at Month 48: number analyzed (Participants) | 2
  Change from Baseline at Month 48 | 1.34 (0.73)
  Change from Baseline at Final Visit: number analyzed (Participants) | 31
  Change from Baseline at Final Visit | 1.91 (1.50)

6. Secondary Outcome: BMI Standard Deviation (SD) Score for Chronological Age Variation
Description: Mean changes of BMI SD score from Pretreatment and from Baseline are reported. SD score is a standard term used in growth studies and represents standard deviations calculated as the patient value minus the mean divided by the SD. SD scores vary depending on the age and sex of the child. It should be noted that only limited patient data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0, 12, 24, 36, 48 and Final Visit (up to 63 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
SD score
  Change from Pretreatment at Baseline: number analyzed (Participants) | 34
  Change from Pretreatment at Baseline | 0.06 (0.27)
  Change from Pretreatment at Month 12: number analyzed (Participants) | 30
  Change from Pretreatment at Month 12 | 0.16 (0.37)
  Change from Pretreatment at Month 24: number analyzed (Participants) | 16
  Change from Pretreatment at Month 24 | -0.01 (0.37)
  Change from Pretreatment at Month 36: number analyzed (Participants) | 3
  Change from Pretreatment at Month 36 | -0.04 (0.63)
  Change from Pretreatment at Month 48: number analyzed (Participants) | 2
  Change from Pretreatment at Month 48 | -0.27 (0.68)
  Change from Pretreatment at Final Visit: number analyzed (Participants) | 31
  Change from Pretreatment at Final Visit | 0.10 (0.46)
  Change from Baseline at Month 12: number analyzed (Participants) | 29
  Change from Baseline at Month 12 | 0.09 (0.27)
  Change from Baseline at Month 24: number analyzed (Participants) | 14
  Change from Baseline at Month 24 | -0.03 (0.27)
  Change from Baseline at Month 36: number analyzed (Participants) | 3
  Change from Baseline at Month 36 | -0.04 (0.38)
  Change from Baseline at Month 48: number analyzed (Participants) | 2
  Change from Baseline at Month 48 | -0.15 (0.45)
  Change from Baseline at Final Visit: number analyzed (Participants) | 31
  Change from Baseline at Final Visit | 0.01 (0.36)

7. Secondary Outcome: Auxological Parameters Variations: Height SD Score
Description: Mean changes of height SD score from Pretreatment and from Baseline are reported. SD score is a standard term used in growth studies and represents standard deviations calculated as the patient value minus the mean divided by the SD. SD scores vary depending on the age and sex of the child. It should be noted that only limited patient data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0, 12, 24, 36, 48 and Final Visit (up to 63 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
SD score
  Change from Pretreatment at Baseline: number analyzed (Participants) | 34
  Change from Pretreatment at Baseline | 0.09 (0.14)
  Change from Pretreatment at Month 12: number analyzed (Participants) | 30
  Change from Pretreatment at Month 12 | -0.05 (0.25)
  Change from Pretreatment at Month 24: number analyzed (Participants) | 16
  Change from Pretreatment at Month 24 | -0.24 (0.43)
  Change from Pretreatment at Month 36: number analyzed (Participants) | 3
  Change from Pretreatment at Month 36 | -0.83 (1.00)
  Change from Pretreatment at Month 48: number analyzed (Participants) | 2
  Change from Pretreatment at Month 48 | -1.68 (0.43)
  Change from Pretreatment at Final Visit: number analyzed (Participants) | 31
  Change from Pretreatment at Final Visit | -0.36 (0.53)
  Change from Baseline at Month 12: number analyzed (Participants) | 29
  Change from Baseline at Month 12 | -0.12 (0.22)
  Change from Baseline at Month 24: number analyzed (Participants) | 14
  Change from Baseline at Month 24 | -0.27 (0.43)
  Change from Baseline at Month 36: number analyzed (Participants) | 3
  Change from Baseline at Month 36 | -0.96 (0.74)
  Change from Baseline at Month 48: number analyzed (Participants) | 2
  Change from Baseline at Month 48 | -1.65 (0.38)
  Change from Baseline at Final Visit: number analyzed (Participants) | 31
  Change from Baseline at Final Visit | -0.43 (0.50)

8. Secondary Outcome: Auxological Parameters Variations: Growth Velocity SD Score
Description: Mean changes of growth velocity SD score from Pretreatment and from Baseline are reported. SD score is a standard term used in growth studies and represents standard deviations calculated as the patient value minus the mean divided by the SD. SD scores vary depending on the age and sex of the child. It should be noted that only limited patient data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0, 12, 24, 36, 48 and Final Visit (up to 63 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
SD score
  Change from Pretreatment at Baseline: number analyzed (Participants) | 26
  Change from Pretreatment at Baseline | -1.85 (2.10)
  Change from Pretreatment at Month 12: number analyzed (Participants) | 24
  Change from Pretreatment at Month 12 | -2.44 (2.08)
  Change from Pretreatment at Month 24: number analyzed (Participants) | 12
  Change from Pretreatment at Month 24 | -3.18 (2.76)
  Change from Pretreatment at Month 36: number analyzed (Participants) | 2
  Change from Pretreatment at Month 36 | -6.97 (5.85)
  Change from Pretreatment at Month 48: number analyzed (Participants) | 2
  Change from Pretreatment at Month 48 | -6.96 (5.79)
  Change from Pretreatment at Final Visit: number analyzed (Participants) | 24
  Change from Pretreatment at Final Visit | -2.70 (2.47)
  Change from Baseline at Month 12: number analyzed (Participants) | 23
  Change from Baseline at Month 12 | -1.06 (1.44)
  Change from Baseline at Month 24: number analyzed (Participants) | 11
  Change from Baseline at Month 24 | -0.92 (1.50)
  Change from Baseline at Month 36: number analyzed (Participants) | 2
  Change from Baseline at Month 36 | -2.79 (1.18)
  Change from Baseline at Month 48: number analyzed (Participants) | 2
  Change from Baseline at Month 48 | -2.65 (1.01)
  Change from Baseline at Final Visit: number analyzed (Participants) | 24
  Change from Baseline at Final Visit | -1.09 (1.30)

9. Secondary Outcome: Auxological Parameters Variations: Weight Variation
Description: Mean changes of weight from Pretreatment and from Baseline are reported. It should be noted that only limited patient data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0, 12, 24, 36, 48 and Final Visit (up to 63 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
kg
  Change from Pretreatment at Baseline: number analyzed (Participants) | 34
  Change from Pretreatment at Baseline | 2.49 (1.53)
  Change from Pretreatment at Month 12: number analyzed (Participants) | 30
  Change from Pretreatment at Month 12 | 7.56 (3.47)
  Change from Pretreatment at Month 24: number analyzed (Participants) | 16
  Change from Pretreatment at Month 24 | 10.13 (4.34)
  Change from Pretreatment at Month 36: number analyzed (Participants) | 3
  Change from Pretreatment at Month 36 | 12.70 (7.05)
  Change from Pretreatment at Month 48: number analyzed (Participants) | 2
  Change from Pretreatment at Month 48 | 12.20 (1.70)
  Change from Pretreatment at Final Visit: number analyzed (Participants) | 31
  Change from Pretreatment at Final Visit | 13.17 (6.21)
  Change from Baseline at Month 12: number analyzed (Participants) | 29
  Change from Baseline at Month 12 | 5.06 (2.79)
  Change from Baseline at Month 24: number analyzed (Participants) | 14
  Change from Baseline at Month 24 | 8.21 (4.17)
  Change from Baseline at Month 36: number analyzed (Participants) | 3
  Change from Baseline at Month 36 | 10.27 (5.11)
  Change from Baseline at Month 48: number analyzed (Participants) | 2
  Change from Baseline at Month 48 | 10.85 (0.92)
  Change from Baseline at Final Visit: number analyzed (Participants) | 31
  Change from Baseline at Final Visit | 10.65 (6.02)

10. Secondary Outcome: Predicted Adult Height SD Score
Description: Mean change of predicted adult height SD score from Pretreatment and from Baseline are reported. SD score is a standard term used in growth studies and represents standard deviations calculated as the patient value minus the mean divided by the SD. SD scores vary depending on the age and sex of the child. It should be noted that only limited patient data was collected after Baseline; all data analysed is presented. Also note that data for this endpoint was analysed for girls only.
Time Frame: Months -6, 0, 12 and Final Visit (up to 63 months)
Population: Analysis performed on female patients in the ITT population, consisting of all enrolled female patients who received at least one injection of study treatment in this follow up study. Only patients with data available at the timepoint of testing are reported.
Measure: Mean (Standard Deviation); unit: SD score
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 34
SD score
  Change from Pretreatment at Baseline: number analyzed (Participants) | 31
  Change from Pretreatment at Baseline | 0.31 (0.18)
  Change from Pretreatment at Month 12: number analyzed (Participants) | 1
  Change from Pretreatment at Month 12 | 0.82 (NA) — No SD is presented since mean value is derived from a single patient
  Change from Pretreatment at Final Visit: number analyzed (Participants) | 4
  Change from Pretreatment at Final Visit | 2.13 (0.87)
  Change from Baseline at Final Visit: number analyzed (Participants) | 4
  Change from Baseline at Final Visit | 1.83 (0.64)

11. Secondary Outcome: Bone Age Maturation
Description: Mean change in difference between bone age and chronological age from Pretreatment and from Baseline are reported. It should be noted that only limited patient data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0 and Final Visit (up to 63 months)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
years
  Change from Pretreatment at Baseline: number analyzed (Participants) | 33
  Change from Pretreatment at Baseline | -0.16 (0.53)
  Change from Pretreatment at Final Visit: number analyzed (Participants) | 5
  Change from Pretreatment at Final Visit | -1.61 (1.04)
  Change from Baseline at Final Visit: number analyzed (Participants) | 5
  Change from Baseline at Final Visit | -1.69 (0.85)

12. Secondary Outcome: Percentage of Girls With a Uterine Length < 36 Millimetres (mm)
Description: Percentage of girls who had a uterine length < 36 mm are reported. It should be noted that only limited patient data was collected after Baseline; all data analysed is presented.
Time Frame: Months -6, 0, 12, 24, 36 and Final Visit (up to 63 months)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 34
percentage of patients
  Pretreatment: number analyzed (Participants) | 33
  Pretreatment | 42.4 [25.48 to 60.78]
  Baseline | 41.2 [24.65 to 59.30]
  Month 12: number analyzed (Participants) | 6
  Month 12 | 16.7 [0.42 to 64.12]
  Month 24: number analyzed (Participants) | 4
  Month 24 | 50.0 [6.76 to 93.24]
  Month 36: number analyzed (Participants) | 1
  Month 36 | 0 [NA to NA] — No CIs are presented since percentage value is derived from a single patient
  Final Visit: number analyzed (Participants) | 4
  Final Visit | 25.0 [0.63 to 80.59]

13. Secondary Outcome: Percentage of Children With a Stabilisation or Regression of Tanner Pubic Hair Pubertal Stage at the End of the Study (Final Visit), Compared to Pretreatment (Month -6) and Baseline (Month 0)
Description: Pubic hair was measured by the Tanner method on a scale of 1 to 6. A low grade (i.e. 1) corresponds to a pre-pubertal stage and a high grade (i.e. 5 or 6) to an adult stage. Percentage of patients who had stabilisation or regression (no change in grade or a reduced grade) of Tanner pubic hair pubertal stage is reported. Study treatment was to last until the end of the therapeutic period; visits for Months 36 and 48 were optional because if the girl was already 11 and the boy already 13, they would have finished the study at a prior visit. The Final Visit was to occur only if the child did not end the study by a complete visit such as at Months 24, 36 or 48. Please also note the additional post-hoc analysis for percentage of children with a stabilisation or regression of Tanner pubic hair pubertal stage which applied the variable Last Visit on Treatment instead of Final Visit.
Time Frame: Months 12, 24, 36, 48 and Final Visit (if applicable; up to 63 months)
Population: Analysis performed on the ITT population, consisting of all enrolled patients who received at least one injection of study treatment in this follow up study.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
percentage of patients
  Compared to Pretreatment (Month -6) | 31.4 [16.85 to 49.29]
  Compared to Baseline (Month 0) | 37.1 [21.47 to 55.08]

14. Post Hoc Outcome: Percentage of Girls With a Stabilisation or Regression of Tanner Breast Pubertal Stage at the End of the Study (Last Visit on Treatment), Compared to Pretreatment (Month -6) and Baseline (Month 0)
Description: One primary efficacy endpoint was to assess efficacy of triptorelin pamoate 11.25 mg with respect to percentage of girls maintaining a regression or stabilisation of sexual maturity (based on Tanner breast pubertal stage) until end of study. Results reported for this primary endpoint applied the variable 'Final Visit' for comparison to Pretreatment and Baseline. Since it was determined that the majority of patients had a Final Visit >3 months after their last injection, a post-hoc analysis of the percentage of girls with regression or stabilisation of Tanner breast pubertal stage was performed which applied the derived variable 'Last Visit on Treatment' to compare to the Pretreatment stage and to Baseline. This post-hoc analysis was judged to be appropriate since triptorelin pamoate 3-month formulation allows release of the active compound over 3 months and beyond this time, pubertal development is expected to progress.
Time Frame: Months 12, 24, 36, 48 and Last Visit on Treatment (if applicable; up to 51 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 34
percentage of patients
  Compared to Pretreatment (Month -6) | 91.2 [76.32 to 98.14]
  Compared to Baseline (Month 0) | 91.2 [76.32 to 98.14]

15. Post Hoc Outcome: Percentage of Children With a Stabilisation or Regression of Tanner Pubic Hair Pubertal Stage at the End of the Study (Last Visit on Treatment), Compared to Pretreatment (Month -6)
Description: One secondary efficacy endpoint in this study was the percentage of children who had stabilisation or regression (no change in grade or a reduced grade) of Tanner pubic hair pubertal stage at the end of the study. Results reported for this secondary endpoint applied the variable 'Final Visit' for comparison to Pretreatment and Baseline. Since it was determined that the majority of patients had a Final Visit >3 months after their last injection, a post-hoc analysis of the percentage of children with regression or stabilisation of Tanner pubic hair pubertal stage was performed which applied the derived variable 'Last Visit on Treatment' for comparison to the Pretreatment stage. This post-hoc analysis was judged to be appropriate since triptorelin pamoate 3-month formulation allows release of the active compound over 3 months and beyond this time, pubertal development is expected to progress.
Time Frame: Months 12, 24, 36, 48 and Last Visit on Treatment (if applicable; up to 51 months)
Population: as for outcome 13
Measure: Number; unit: percentage of patients
Arm/Group | Triptorelin Pamoate 11.25 mg
Number analyzed (Participants) | 35
percentage of patients | 57.1

ADVERSE EVENTS:
Time Frame: Up to 51 months (up to 48 months treatment + 3 months follow up)
Description: Adverse event (AE) data is reported as treatment-emergent AEs
Arm/Group | Triptorelin Pamoate 11.25 mg
Serious Adverse Events (participants affected / at risk) | 3/35
Other Adverse Events (participants affected / at risk) | 16/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate 11.25 mg (N=35)
Gait disturbance (General disorders) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate 11.25 mg (N=35)
Abdominal pain (Gastrointestinal disorders) | 6 (9)
Vomiting (Gastrointestinal disorders) | 2 (2)
Injection site pain (General disorders) | 4 (6)
Insomnia (Psychiatric disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 2 (2)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Hot flush (Vascular disorders) | 3 (3)
Weight increased (Investigations) | 2 (2)

LIMITATIONS AND CAVEATS:
Since almost no hormonal data was collected after Baseline and only limited data was collected after Baseline for all other efficacy endpoints, only limited post-Baseline data is reported for the trial overall. All data analysed has been presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days